CLINICAL TRIAL: NCT03031626
Title: Comparison of Therapeutic Oxygen Versus Medical Air for the Treatment of Central Sleep Apnea in Infants and Children With Prader Willi Syndrome: A Proof of Concept Study
Brief Title: Oxygen Versus Medical Air for Treatment of CSA in Prader Will Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Respirologist, Clinician Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000053577
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Sleep Apnea, Central; Prader-Willi Syndrome
MeSH Terms: conditions — Sleep Apnea, Central; Prader-Willi Syndrome

STUDY DESIGN:
Intervention Model Description: The screening visit will occur during a regularly scheduled clinic visit. The patients that have consented for the study will all undergo the baseline PSG. Only patients with clinically significant CSA after Visit 1 will undergo randomization and complete Visit 2.
  Those who have a CAHI greater or equal to 5 will be randomly assigned to Arm A or Arm B. Randomization will be performed using a computer with random numbers drawn. Arm A will receive Medical Air followed by Oxygen and Arm B will receive Oxygen followed by Medical Air.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The split-night polysomnograms (Arm A, Arm B) will be scored by a blinded independent sleep technologist. A Sleep Physician will report the sleep study and be blinded as to the gas assignment (ie Arm A or Arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Medical air followed by oxygen (Experimental)
  Interventions: Biological: Medical Air vs Oxygen
- Arm B: Oxygen followed by medical air (Experimental)
  Interventions: Biological: Medical Air vs Oxygen

INTERVENTIONS:
Biological: Medical Air vs Oxygen — Medical Air/Oxygen will be given

SUMMARY:
The aim of this study is to determine if treatment with Medical Air (21% oxygen in room air) compared to supplemental oxygen (100% oxygen) will lead to similar improvements in the central apnea-hypopnea index (CAHI) for infants with Prader-Willi Syndrome.

Despite the vast amount of research investigating the cause of central sleep apnea, there remain gaps in knowledge, lending to further research efforts. The decision to compare oxygen to medical air is based on several theorized mechanisms. The first of which is the supposition that provision of medical air may act as an arousal stimulus for the hypothalamus, thereby preventing sleep disordered breathing. Secondly, the hypercapnic challenge performed by Livingston et al demonstrated a delayed hypercapneic arousal response in PWS subjects despite simultaneous hyperoxia, leading us to question if therapeutic oxygen really plays a significant role in treating CSA. Lastly, the delivery of medical air via nasal prongs may provide sufficient arousal to terminate the cycle of events leading to central apnea, as described by Urquhart et al.

A deeper understanding of central sleep apnea is essential to ameliorating its adverse sequelae, which include symptoms of ADHD, impaired attention, behavioral problems, and academic difficulties.

ELIGIBILITY:
Inclusion Criteria:

1. infants under age two with genetically confirmed Prader-Willi Syndrome
2. referred to HSC sleep clinic for evaluation with polysomnogram prior to initiation of growth hormone
3. infants found to have clinically significant central sleep apnea, defined as an apnea-hypopnea index (AHI) equal to or greater than 5

Exclusion Criteria:

1. infants delivered prematurely (less than 37 weeks gestational age)
2. term infants with a history of hypoxic-ischemic encephalopathy or stroke
3. any concurrent diagnoses that may cause sleep-disordered breathing (ie. craniofacial abnormalities, arnold-chiari malformation, etc)
4. infants with a need for daytime supplemental oxygen (ie. cardiac anomalies)
5. infants found to have low baseline oxygen saturations on PSG

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Delta CAHI1 | 2 years
  Difference in CAHI at baseline compared to supplemental oxygen Delta CAHI1: CAHIoxygen - CAHIbaseline
Delta CAHI2 | 2 years
  Difference in CAHI at baseline compared to medical air Delta CAHI2: CAHImedical air - CAHIbaseline
Difference in CAHI1 and CAHI2 | 2 years
  A comparison of change in CAHI1 and change in CAHI2 DeltaCAHI1: DeltaCAHI2

SECONDARY OUTCOMES:
Arousal Index1 | 2 years
  Difference in Arousal Index at baseline compared to medical air Delta Arousal Index: Arousal Indexmedical air - Arousal Indexbaseline
Arousal Index2 | 2 years
  Difference in Arousal Index at baseline compared to Supplemental oxygen Delta Arousal Index: Arousal Indexoxygen - Arousal Indexbaseline
Desaturation Index1 | 2 years
  Difference in Desaturation Index at baseline compared to medical air Delta Arousal Index: Desaturation Indexmedical air - Desaturation Indexbaseline
Desaturation Index2 | 2 years
  Difference in Desaturation Index at baseline compared to supplemental oxygen Delta Arousal Index: Desaturation Indexoxygen - Desaturation Indexbaseline

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided